CLINICAL TRIAL: NCT02122445
Title: Effectiveness of Cramer Sports Motion Tape on Low Back Pain Patients' Pain and Muscle Activation
Brief Title: Cramer Sports Motion Tape and Low Back Pain EMG
Acronym: KT_LBP_EMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sport and Spine Rehab Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSR03
Record Dates: First submitted 2014-04-21; First posted 2014-04-24 (Estimated); Results first posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-01

CONDITIONS: Low Back Pain
Keywords: Gluteus Maximum; Gluteus Medius; TFL; EMG; Flexion-Response Phenomenon; Thera-Band; kinesiology tape
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low Back Pain (Experimental): Lower body exercises before and after the application of Cramer Sports Motion tape
  Interventions: Device: Cramer Sports Motion Tape

INTERVENTIONS:
Device: Cramer Sports Motion Tape — lower body exercises with and without Cramer Sports Motion tape applied to the hip

SUMMARY:
Low back pain is a problem which affects up to 70-80% of people in their lifetime. In the United States, it is estimated that the total direct and indirect costs of low back pain combined ranges from $19.6 to $118.8 billion. Recent studies have shown the importance of the gluteal musculature in the treatment of low back pain. It was found that the gluteus maximus (Gmax) is significantly more active in a low back pain population compared to a healthy population, indicating the low back pain population relied on the Gmax to fire more to overcome the gluteal weakness. A new approach to treating musculoskeletal conditions is a taping technique designed to target muscles and lymphatic system. Limited research is available for the treatment of specific conditions, including low back pain, but it is theorized to inhibit or facilitate the muscle, improve blood flow, reduce pain, and improve joint alignment. Methods: The purpose of this study is to determine the immediate and delayed effectiveness of Cramer® Sports Motion Tape on Gmax and lumbar paraspinal activation in a chronic mechanical low back pain population. A convenience sample of 20 new patients with current, chronic low back pain, no current neurologic signs or symptoms, no previous spinal surgery, no corticosteroid treatment within the last two weeks, and who are not pregnant will be recruited for this study. Patients will sign an informed consent, complete all initial paperwork. Surface electromyography will be used to quantify the activity level of the Gmax and lumbar paraspinals (LP). The MVIC will be estimated for each muscle group and the patient will perform a series of 4 randomized exercises, 5 repetitions each; Clams with Resistance, Standing Hip Abduction with Resistance, Sidelying Hip Abduction, and a forward bend. After each exercise the patient will rate "How hard they are working" on the RISE scale. Following the initial test, Cramer® Sports Motion Tape will be applied to the gluteal and low back area. After the tape is applied, the EMG exercise protocol will be repeated. The tape will be left on until the patient returns for their next appointment, within 24 to 48 hours, where they will have a delayed post-test. Patients will rate their pain, surface electrodes will be applied to the previous testing sites, and MVIC will be retested for each muscle group. The patient will perform the same protocol that was performed in the initial testing session. The EMG signals will be smoothed, rectified and analyzed using a root-mean-square algorithm. The investigators will use visual onset and offset of the EMG signal amplitude to select the middle 3 trials. Average activation and peak activation will be determined and compared to the MVIC for each muscle group, and expressed as a %MVIC. This will allow %MVIC to be compared and rank order among groups and muscles.

ELIGIBILITY:
Inclusion Criteria:

* must be recruited within the first 2 to 3 therapy visits
* have a diagnosis of chronic mechanical low back pain
* 18-65

Exclusion Criteria:

* no current neurologic signs or symptoms
* no previous spinal surgery
* no corticosteroid treatment within the last two weeks
* may not be pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barton Bishop, DPT, Principal Investigator — Sport & Spine Rehab Clinical Research Foundation
Locations (1):
- Sport & Spine Rehab, Rockville, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Low back pain patients, evaluated within the first 2 initial visits of treatment at an outpatient rehabilitation clinic.
Period: Overall Study
Arm/Group | Low Back Pain
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Low Back Pain
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 40.05 [19 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Percent of Maximal Voluntary Isometric Contraction (%MVIC)
Description: 3 muscles during 4 exercises (ClamsR, Sidelying, StandingAB, ForwardBend) at 3 time points (Baseline[T1], Immediate post[T2], 24hrs[T3]), were analyzed in 20 subjects, totaling 720 data points. Maximal voluntary isometric contraction(MVIC) was assessed using the standard manual muscle testing positions. For each subject, the EMG signals of the muscles during the exercises were smoothed, rectified and analyzed using a root-mean-square algorithm and the greatest activation of each muscle was used. After the peak activation(PA) for each muscle was determined, it was compared to the MVIC of the reference exercise for the respective muscle group, and expressed as a percent of MVIC (%MVIC). In some cases the %MVIC is greater than 100% because the MVIC was assessed during a manual muscle test position. During an exercise some muscles generated greater PA and therefore when calculated the %MVIC was greater than 100%. Due to the amount of data, we have provided the Gmax %MVIC results.
Time Frame: % Maximal Voluntary Isometric Contracion (%MVIC)
Measure: Mean (Full Range); unit: % of Max Voluntary Isometric Contraction
Arm/Group | Low Back Pain
Number analyzed (Participants) | 20
% of Max Voluntary Isometric Contraction
  ClamsR Gmax T1 | 226.41 [27.18 to 544.47]
  ClamsR Gmax T2 | 250.51 [39.28 to 1096.71]
  ClamsR Gmax T3 | 162.47 [15.15 to 938.65]
  Sidelying Gmax T1 | 205.82 [22.98 to 1253.38]
  Sidelying Gmax T2 | 176.24 [16.54 to 895.55]
  Sidelying Gmax T3 | 139.20 [14.13 to 668.71]
  StandingAB Gmax T1 | 196.31 [29.82 to 1057.82]
  StandingAB Gmax T2 | 186.15 [26.36 to 750]
  StandingAB Gmax T3 | 124.84 [35.25 to 550.10]
  ForwardBend Gmax T1 | 54.34 [24.64 to 127.10]
  ForwardBend Gmax T2 | 55.57 [19.78 to 167.64]
  ForwardBend Gmax T3 | 52.05 [11.86 to 123.36]

2. Secondary Outcome: Perceived Exertion
Description: The amount of perceived exertion was reported for each of the 4 exercises (ClamsR, Sidelying, StandingAB, ForwardBend) at 3 time points (Baseline[T1], Immediate post[T2], 24hrs[T3]), by 20 subjects, totaling 240 data points. This was measured using the TheraBand(R) Resistance Intensity Scale for Exercise (RISE Scale). Participants were asked to rate their perceived exertion on a scale of 0 to 10, 0 being no resistance and 10 being maximum resistance. The results of the 20 subjects were averaged for each exercise at each time point.
Time Frame: Perceived Exertion
Measure: Mean (Full Range); unit: units on a scale, from 0 to 10
Arm/Group | Low Back Pain
Number analyzed (Participants) | 20
units on a scale, from 0 to 10
  Clams T1 | 2.95 [0 to 5]
  Clams T2 | 2.6 [0 to 5]
  Clams T3 | 2.55 [0 to 6]
  Sidelying T1 | 2.75 [1 to 6]
  Sidelying T2 | 2.15 [0 to 5]
  Sidelying T3 | 2.15 [0 to 5]
  StandingAB T1 | 3.1 [0 to 6]
  StandingAB T2 | 2.5 [0 to 7]
  StandingAB T3 | 2.4 [0 to 6]
  ForwardBend T1 | 3.5 [0 to 8]
  ForwardBend T2 | 2.3 [0 to 8]
  ForwardBend T3 | 2.5 [0 to 6]

ADVERSE EVENTS:
Arm/Group | Low Back Pain
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No